CLINICAL TRIAL: NCT07338032
Title: Task Specific Training and Conventional Physical Therapy on Ankle Dorsiflexion in Sub-acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Rimsha Khalid, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/0040
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Subacute Stroke
Keywords: Ankle Dorsiflexion; Gait; Stroke Rehabilitation; Task-Specific Training; Time Up and Go Test
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-Specific Training + Conventional Physiotherapy (Experimental): Participants will receive an 8-week program (3 sessions/week; ~45 min/session) consisting of task-specific gait and ankle-focused functional activities combined with conventional physiotherapy. Task-specific training includes goal-directed walking tasks (forward, backward, and sideways walking with therapist guarding; structured sets and rest). Additional task-oriented exercises may include toe walking, heel raises on a step, single-leg stance on a foam surface, active toe lifts, and resisted ankle dorsiflexion using weighted boots or resistance bands. Conventional components (as per protocol) may be provided alongside to support strength, flexibility, and safe gait practice.
  Interventions: Behavioral: Task-Specific Training Combined With Conventional Physiotherapy
- Conventional Physiotherapy (Ankle Dorsiflexor Strengthening) (Other): Participants will receive conventional physiotherapy for 8 weeks (3 sessions/week; ~45-60 min/session) focusing on ankle dorsiflexor strengthening and flexibility. The strengthening program includes isometric ankle dorsiflexion against manual resistance (held contractions with rest intervals, repeated in sets) and progressive concentric dorsiflexion strengthening using resistance bands or ankle weights with gradual progression in intensity and repetitions across the intervention period. Plantarflexor stretching will be performed as part of the protocol (held stretches repeated per session). The program is delivered by an experienced physiotherapist under standardized safety and positioning instructions.
  Interventions: Behavioral: Conventional Physiotherapy for Ankle Dorsiflexor Strengthening

INTERVENTIONS:
Behavioral: Task-Specific Training Combined With Conventional Physiotherapy — This intervention consists of task-specific training combined with conventional physiotherapy delivered over 8 weeks, with three supervised sessions per week (approximately 45 minutes per session). Task-specific training emphasizes repetitive, goal-directed functional activities designed to enhance ankle dorsiflexion during gait. Exercises include forward, backward, and sideways walking under therapist supervision, toe walking, heel raises on a step, single-leg stance tasks, active toe lifts, and resisted ankle dorsiflexion using weighted boots or resistance bands. Conventional physiotherapy components, including strengthening and flexibility exercises for the ankle dorsiflexors, may be incorporated alongside task-oriented activities as per protocol. All sessions are delivered by a qualified physiotherapist following standardized safety and progression guidelines.
  Arms: Task-Specific Training + Conventional Physiotherapy
Behavioral: Conventional Physiotherapy for Ankle Dorsiflexor Strengthening — This intervention consists of a conventional physiotherapy program focused on ankle dorsiflexor strengthening and flexibility, delivered over 8 weeks with three supervised sessions per week (45-60 minutes per session). The program includes isometric ankle dorsiflexion exercises against manual resistance, held contractions with rest intervals, and progressive concentric dorsiflexion strengthening using resistance bands or ankle weights with gradual increases in intensity and repetitions. Passive and active stretching of the plantarflexor muscles is also included. All exercises are administered by an experienced physiotherapist using standardized positioning, safety precautions, and progression criteria.
  Arms: Conventional Physiotherapy (Ankle Dorsiflexor Strengthening)

SUMMARY:
This study is a randomized clinical trial designed to compare two physiotherapy rehabilitation approaches for people in the sub-acute phase after stroke (2-6 months after stroke). Stroke often causes weakness of the ankle dorsiflexor muscles, which can lead to foot drop and difficulty walking safely. Improving ankle control may help balance and functional mobility.

Eligible participants will be recruited from two tertiary care hospitals using purposive sampling and enrolled after providing informed consent. After baseline assessment, participants will be randomly allocated to one of two groups. The experimental group will receive task-specific training combined with conventional physiotherapy, and the control group will receive conventional physiotherapy alone. Treatment will be delivered for 8 weeks, three sessions per week.

Outcomes will be assessed at baseline and after completion of the 8-week intervention. The primary outcomes are ankle dorsiflexor strength measured by Manual Muscle Testing (MMT) and functional mobility measured by the Timed Up and Go (TUG) test. Balance measured by the Berg Balance Scale (BBS) is the secondary outcome. An independent outcome assessor who is not involved in treatment delivery will conduct the assessments to reduce measurement bias.

DETAILED DESCRIPTION:
This interventional randomized clinical trial will be conducted over nine months following institutional ethical approval at the University of Lahore Teaching Hospital, Lahore, and Sharif City Medical Hospital. Participants will be recruited using a non-probability purposive sampling technique from the study settings. Eligibility criteria include adults aged 40-65 years with sub-acute stroke (2-6 months post-stroke), ability to walk with or without an assistive device, minimum ankle plantarflexion-dorsiflexion range, ability to follow commands (MMSE ≥24), and plantarflexor spasticity grade 1 or 1+. Key exclusions include uncorrected sensory impairment, neglect, aphasia, painful musculoskeletal conditions, other neurological disorders, and concurrent participation in other rehabilitation programs.

After written informed consent, participants will undergo baseline assessment of functional mobility, balance, and ankle dorsiflexor strength. Randomization will be performed after enrollment using an online randomization tool, with allocation concealment implemented through a sealed-envelope method. This study will use a single-blinded approach in which outcome assessment is conducted by an independent assessor who is not involved in treatment delivery and is unaware of group allocation.

Participants will be allocated to one of two parallel groups:

Group A (Experimental): Task-specific training plus conventional physiotherapy Participants will receive an 8-week program, three sessions per week, approximately 45 minutes per session. Task-specific gait training will include functional walking activities (forward, backward, and sideways walking with appropriate safety guarding and rest intervals). Additional task-oriented lower-limb activities may include toe walking, heel raises on a step, single-leg stance tasks, active toe lifts, and resisted ankle dorsiflexion exercises. Conventional physiotherapy components may be provided alongside task-specific training as per protocol.

Group B (Control): Conventional physiotherapy only Participants will receive an 8-week conventional physiotherapy program, three sessions per week (approximately 45-60 minutes/session), focusing on ankle dorsiflexor strengthening and flexibility. The program will include isometric dorsiflexion against resistance, progressive concentric dorsiflexion strengthening using bands/weights with planned progression, and plantarflexor stretching.

Outcome Measures and Time Points Assessments will be performed at baseline and immediately post-intervention (after 8 weeks). Primary outcomes are (1) ankle dorsiflexor strength assessed by Manual Muscle Testing (MMT) and (2) functional mobility assessed by the Timed Up and Go (TUG) test. Secondary outcome is balance assessed by the Berg Balance Scale (BBS). Data will be analyzed using SPSS with significance level set at p < 0.05.

Sample Size Sample size was calculated using Epitool as 54 participants (27 per group). To account for an anticipated 20% dropout rate, the target enrollment will be 66 participants (33 per group).

ELIGIBILITY:
Inclusion Criteria:

* Onset of stroke 2-6 months before study enrollment (Van Criekinge et al., 2022).
* Ability to walk with or without an assistive device (Khallaf, 2020).
* Presence of a minimum of 8-10 Degree of ankle plantarflexion-dorsiflexion range
* Ability to follow a three-step command, MMSE 24 (Srivastava et al., 2024).
* Spasticity of plantarflexers 1 or 1+ (Abd Elsabour et al., 2025).
* Not participating in any other form of physical rehabilitation. No lumber radiculopathy (Srivastava et al., 2024).

Exclusion Criteria:

* Uncorrected vision and hearing loss or sensory impairment (Van Criekinge et al., 2022).
* Unilateral or Visual neglect (Van Criekinge et al., 2022).
* Sensory or global aphasia (Khallaf, 2020).
* Pain or musculoskeletal or any other neurological disorder (Srivastava et al., 2024).
* Carcinoma (Srivastava et al., 2024).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-01-03 (Actual)

PRIMARY OUTCOMES:
Ankle Dorsiflexor Muscle Strength | Baseline (pre-intervention) and immediately after completion of the 8-week intervention program
  Ankle dorsiflexor muscle strength will be assessed using Manual Muscle Testing (MMT). Muscle strength is graded on a standardized ordinal scale ranging from 0 (no visible or palpable muscle contraction) to 5 (normal muscle strength against full resistance). MMT will be performed by a trained assessor using standardized positioning and resistance techniques to ensure consistency. The assessment focuses on the affected lower limb ankle dorsiflexor muscles, which are essential for foot clearance and gait during walking.
Functional Mobility Assessed by the Timed Up and Go Test | Baseline (pre-intervention) and immediately after completion of the 8-week intervention program
  Functional mobility will be evaluated using the Timed Up and Go (TUG) test. The test measures the time, in seconds, required for a participant to stand up from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down. Lower completion times indicate better functional mobility. The TUG test will be administered under standardized conditions by a trained assessor to ensure reliability and reproducibility.

SECONDARY OUTCOMES:
Balance Assessed by the Berg Balance Scale | Baseline (pre-intervention) and immediately after completion of the 8-week intervention program
  Balance will be assessed using the Berg Balance Scale (BBS), a validated clinical tool consisting of 14 functional balance tasks such as sitting, standing, transfers, reaching, turning, and single-leg stance. Each task is scored on a 5-point ordinal scale (0-4), with a maximum total score of 56. Higher scores indicate better balance performance. The BBS will be administered by a trained assessor following standardized instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorsch, S., Ada, L., Canning, C. G., & Al-Zoubi, F. (2023). Bobath therapy is inferior to task-specific training and not superior to usual care after stroke: A systematic review. Journal of NeuroEngineering and Rehabilitation, 20, 12. https://doi.org/10.1186/s12984-023-01154-6
- [Background] Belghith K, Zidi M, Vincent L, Fedele JM, Bou-Serhal R, Maktouf W. Eccentric strengthening vs. conventional therapy in sub-acute stroke survivors: a randomized controlled trial. Front Neurol. 2025 Jan 23;15:1398860. doi: 10.3389/fneur.2024.1398860. eCollection 2024. PMID 39917437